CLINICAL TRIAL: NCT00736775
Title: A Phase I, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Intravenous MABT5102A Administered in a Single-Dose, Dose-Escalation Stage Followed by a Multidose, Parallel-Treatment Stage in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: A Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Anti-Abeta (MABT5102A) in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Disclosures Group, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABE4427g
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: Alzheimer's Disease
Keywords: AD; Alzheimer's; Alzheimers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: anti-Abeta — Intravenous single and multiple doses
Drug: placebo — Intravenous single and multiple doses

SUMMARY:
This is a Phase I, multicenter, randomized, double-blind, placebo-controlled study that will be conducted in the United States and consists of a single ascending-dose stage followed by a multidose, parallel-treatment stage. This study will be conducted in approximately 50 adult patients between 50-85 years old who have mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD according to the NINCDS-ADRDA Criteria
* Approved AD treatments (AchE inhibitors+/-memantine) must be stable for ≥ 3 months prior to screening
* Other prescription medications must be stable for ≥ 1 month prior to screening

Exclusion Criteria:

* Female patients with reproductive potential
* History or presence of any clinically significant CNS disease
* History of treatment with any protein therapeutic targeting Abeta

Ages: 50 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple doses of MABT5102A | Through study completion or early study discontinuation

SECONDARY OUTCOMES:
Pharmacokinetics of MABT5102A after single and multiple doses | Through study completion or early study discontinuation
Immunogenicity of MABT5102A after single and multiple doses | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Carole Ho, M.D., Study Director — Genentech, Inc.